CLINICAL TRIAL: NCT03675399
Title: Effect of Isometric Exercise on Pain Perception in Subjects With Rotator Cuff Related Shoulder Pain
Brief Title: Effect of Isometric Exercise on Pain Perception in Rotator Cuff Related Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Mercè Balasch i Bernat, PhD Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1528701290644
Record Dates: First submitted 2018-09-13; First posted 2018-09-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Rotator Cuff Tendinitis
Keywords: isometric exercise; rotator cuff; pain threshold
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Exercise sessions were delivered by a physiotherapist who was not involved in the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supra-threshold isometric exercise (Experimental): Participants will perform 10 isometric external rotation supra-threshold contractions of the affected shoulder, each held for 15 seconds, with resting intervals of 15 seconds between contractions.
  Interventions: Other: Supra-threshold isometric exercise
- Infra-threshold isometric exercise (Experimental): Participants will perform 10 isometric external rotation infra-threshold contractions of the affected shoulder, each held for 15 seconds, with resting intervals of 15 seconds between contractions.
  Interventions: Other: Infra-threshold isometric exercise
- Control (No Intervention): Participants will remain resting.

INTERVENTIONS:
Other: Supra-threshold isometric exercise — The supra-threshold intensity will be stablished at 120% of participant's PFIS pre-session measurement (20% above the individual's pain threshold).
  Arms: Supra-threshold isometric exercise
Other: Infra-threshold isometric exercise — The infra-threshold intensity will be stablished at 80% of participant's PFIS pre-session measurement (20% bellow the individual's pain threshold).
  Arms: Infra-threshold isometric exercise

SUMMARY:
The aim of this study is to compare the immediate effects of an acute bout of isometric exercise of the shoulder external rotator muscles above and below pain threshold on pain intensity, pain threshold, conditioned pain modulation and pain free force in external rotation. To evaluate the results of the exercise, the subjects will be assessed at pre-intervention, immediately post-intervention and after and 45 minutes after each experimental condition.

DETAILED DESCRIPTION:
The aim of this study is to compare the immediate effects of an acute bout of isometric exercise of the shoulder external rotator muscles above and below pain threshold on pain intensity, pain threshold, conditioned pain modulation and pain free force in external rotation.

It will consist of a randomized three-treatment parallel-design study. The sample will consist of subjects with rotator cuff related shoulder pain (RCRSP). Once the sample is selected, subjects will participate in three experimental sessions, which will occur in a randomized order: two exercise sessions (supra-threshold and infra-threshold isometric exercise) and one control session. In the first session, information regarding clinical and demographical aspects will be collected. A washout period of approximately 48 hours will separate each of the experimental sessions.

To evaluate the results of the exercise, the subjects will be assessed at pre-intervention, immediately post-intervention and 45 minutes after each experimental condition. Pain intensity, Pressure Pain Thresholds (PPT), Conditioned Pain Modulation (CPM), maximal voluntary isometric contraction (MVIC) and pain free isometric strength (PFIS) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years (likelihood of patients > 80 having degenerative changes in the shoulder is increased)
* pain localised to the proximal anterolateral shoulder region
* positive for pain on at least one of the following three impingement tests: Hawkins-Kennedy, Neer's, Jobe's
* positive for pain on resisted external rotation and/or abduction.

Exclusion Criteria:

* shoulder surgery within last 6 months
* reasons to suspect systemic pathology including inflammatory disorders, cervical repeated movement testing affects shoulder pain and/or range of movement, passive external rotation deficit greater (less than 30º or a range of motion reduction of 50% or more as compared to the contralateral side), upper limb tension test A for cervical radiculopathy
* atraumatic degenerative rotator cuff tear based on the cluster of clinical tests (painful arc, drop arm test, and marked weakness into ER all three positive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain).
Pain intensity | Immediately post-intervention
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain).
Pain intensity | 45 minutes post-intervention
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Lower values represent a better outcome (less pain).

SECONDARY OUTCOMES:
Pressure Pain Thresholds (PPT) | Baseline, immediately post-intervention and 45 minutes post-intervention
  PPTs will be recorded using an electronic algometer at the ipsilateral m. infraspinatus, the contralateral resting m. infraspinatus and the contralateral resting m. quadriceps. Higher values represent a better outcome.
Pressure Pain Thresholds (PPT) | Immediately post-intervention
  PPTs will be recorded using an electronic algometer at the ipsilateral m. infraspinatus, the contralateral resting m. infraspinatus and the contralateral resting m. quadriceps. Higher values represent a better outcome.
Pressure Pain Thresholds (PPT) | 45 minutes post-intervention
  PPTs will be recorded using an electronic algometer at the ipsilateral m. infraspinatus, the contralateral resting m. infraspinatus and the contralateral resting m. quadriceps. Higher values represent a better outcome.
Conditioned pain modulation (CPM) | Baseline
  CPM will be tested using the upper extremity submaximal effort tourniquet test.
Conditioned pain modulation (CPM) | Immediately post-intervention
  CPM will be tested using the upper extremity submaximal effort tourniquet test.
Conditioned pain modulation (CPM) | 45 minutes post-intervention
  CPM will be tested using the upper extremity submaximal effort tourniquet test.
Maximal voluntary isometric contraction (MVIC) | Baseline
  MVIC will be measured at both m. infraspinatus and m. quadriceps of the non-affected side using a digital force gauge.
Maximal voluntary isometric contraction (MVIC) | Immediately post-intervention and 45 minutes post-intervention
  MVIC will be measured at both m. infraspinatus and m. quadriceps of the non-affected side using a digital force gauge.
Maximal voluntary isometric contraction (MVIC) | 45 minutes post-intervention
  MVIC will be measured at both m. infraspinatus and m. quadriceps of the non-affected side using a digital force gauge.
Pain free isometric strength/threshold (PFIS) | Baseline
  PFIS will be assessed at m. infraspinatus of the affected shoulder
Pain free isometric strength/threshold (PFIS) | Immediately post-intervention
  PFIS will be assessed at m. infraspinatus of the affected shoulder
Pain free isometric strength/threshold (PFIS) | 45 minutes post-intervention
  PFIS will be assessed at m. infraspinatus of the affected shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Mercè Balasch i Bernat, PhD, Principal Investigator — Universitat de València
Locations (2):
- Spain (2):
  - Mercè Balasch i Bernat, Valencia, Valencia
  - Mercè Balasch i Bernat, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Watts AR, Williams B, Kim SW, Bramwell DC, Krishnan J. Shoulder impingement syndrome: a systematic review of clinical trial participant selection criteria. Shoulder Elbow. 2017 Jan;9(1):31-41. doi: 10.1177/1758573216663201. Epub 2016 Aug 20. PMID 28572848
- [Background] Maenhout AG, Mahieu NN, De Muynck M, De Wilde LF, Cools AM. Does adding heavy load eccentric training to rehabilitation of patients with unilateral subacromial impingement result in better outcome? A randomized, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1158-67. doi: 10.1007/s00167-012-2012-8. Epub 2012 May 12. PMID 22581193
- [Result] Luime JJ, Koes BW, Miedem HS, Verhaar JA, Burdorf A. High incidence and recurrence of shoulder and neck pain in nursing home employees was demonstrated during a 2-year follow-up. J Clin Epidemiol. 2005 Apr;58(4):407-13. doi: 10.1016/j.jclinepi.2004.01.022. PMID 15862727
- [Result] Lewis J. Rotator cuff related shoulder pain: Assessment, management and uncertainties. Man Ther. 2016 Jun;23:57-68. doi: 10.1016/j.math.2016.03.009. Epub 2016 Mar 26. PMID 27083390
- [Result] Littlewood C, Malliaras P, Chance-Larsen K. Therapeutic exercise for rotator cuff tendinopathy: a systematic review of contextual factors and prescription parameters. Int J Rehabil Res. 2015 Jun;38(2):95-106. doi: 10.1097/MRR.0000000000000113. PMID 25715230
- [Result] Littlewood C, Ashton J, Chance-Larsen K, May S, Sturrock B. Exercise for rotator cuff tendinopathy: a systematic review. Physiotherapy. 2012 Jun;98(2):101-9. doi: 10.1016/j.physio.2011.08.002. Epub 2011 Oct 5. PMID 22507359
- [Result] Smith BE, Hendrick P, Smith TO, Bateman M, Moffatt F, Rathleff MS, Selfe J, Logan P. Should exercises be painful in the management of chronic musculoskeletal pain? A systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(23):1679-1687. doi: 10.1136/bjsports-2016-097383. Epub 2017 Jun 8. PMID 28596288
- [Result] Holmgren T, Bjornsson Hallgren H, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. BMJ. 2012 Feb 20;344:e787. doi: 10.1136/bmj.e787. PMID 22349588
- [Result] Littlewood C, Bateman M, Brown K, Bury J, Mawson S, May S, Walters SJ. A self-managed single exercise programme versus usual physiotherapy treatment for rotator cuff tendinopathy: a randomised controlled trial (the SELF study). Clin Rehabil. 2016 Jul;30(7):686-96. doi: 10.1177/0269215515593784. Epub 2015 Jul 9. PMID 26160149
- [Result] Coombes BK, Wiebusch M, Heales L, Stephenson A, Vicenzino B. Isometric Exercise Above but not Below an Individual's Pain Threshold Influences Pain Perception in People With Lateral Epicondylalgia. Clin J Pain. 2016 Dec;32(12):1069-1075. doi: 10.1097/AJP.0000000000000365. PMID 26889612
- [Result] Naugle KM, Fillingim RB, Riley JL 3rd. A meta-analytic review of the hypoalgesic effects of exercise. J Pain. 2012 Dec;13(12):1139-50. doi: 10.1016/j.jpain.2012.09.006. Epub 2012 Nov 8. PMID 23141188
- [Result] Rio E, Kidgell D, Purdam C, Gaida J, Moseley GL, Pearce AJ, Cook J. Isometric exercise induces analgesia and reduces inhibition in patellar tendinopathy. Br J Sports Med. 2015 Oct;49(19):1277-83. doi: 10.1136/bjsports-2014-094386. Epub 2015 May 15. PMID 25979840
- [Derived] Balasch-Bernat M, Lluch E, Vaegter HB, Duenas L. Should Exercises be Painful or not? Effects on Clinical and Experimental Pain in Individuals with Shoulder Pain. J Pain. 2021 Oct;22(10):1246-1255. doi: 10.1016/j.jpain.2021.03.153. Epub 2021 Apr 20. PMID 33887445